CLINICAL TRIAL: NCT05478525
Title: A Phase 2 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Safety, Tolerability, and Pharmacodynamic Effects of GLY-200 in Type 2 Diabetic Patients
Brief Title: A Study Evaluating the Safety, Tolerability, and Pharmacodynamic Effects of GLY-200 in Type 2 Diabetic Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Glyscend, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GLY-200-02
Record Dates: First submitted 2022-07-26; First posted 2022-07-28 (Actual); Results first posted 2025-02-10 (Actual); Last update posted 2025-02-10 (Actual); Status verified 2025-02

CONDITIONS: Type 2 Diabetes
Keywords: Type 2 Diabetes; Diabetes Mellitus, Type 2; GLY-200; Glyscend, Inc.
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- 0.5 g GLY-200 (Experimental): 0.5 g GLY-200 (1 x 0.5 g capsule) twice a day (BID)
  Interventions: Drug: GLY-200
- 1.0 g GLY-200 (Experimental): 1.0 g GLY-200 (2 x 0.5 g capsule) twice a day (BID)
  Interventions: Drug: GLY-200
- 2.0 g GLY-200 (Experimental): 2.0 g GLY-200 (4 x 0.5 g capsule) twice a day (BID)
  Interventions: Drug: GLY-200
- Placebo for 0.5 g GLY-200 arm (Placebo Comparator): 1 placebo capsule twice a day (BID)
  Interventions: Drug: Placebo
- Placebo for 1.0 g GLY-200 arm (Placebo Comparator): 2 placebo capsules twice a day (BID)
  Interventions: Drug: Placebo
- Placebo for 2.0 GLY-200 arm (Placebo Comparator): 4 placebo capsules twice a day (BID)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: GLY-200 — 0.5 g GLY-200 (1 x 0.5 g capsule) BID for 14 days (n=12)
  Arms: 0.5 g GLY-200
Drug: GLY-200 — 1.0 g GLY-200 (2 x 0.5 g capsules) BID for 14 days (n=12)
  Arms: 1.0 g GLY-200
Drug: GLY-200 — 2.0 g GLY-200 (4 x 0.5 g capsules) BID for 14 days (n=12)
  Arms: 2.0 g GLY-200
Drug: Placebo — 1 placebo capsule BID for 14 days (n=4)
  Arms: Placebo for 0.5 g GLY-200 arm
Drug: Placebo — 2 placebo capsules BID for 14 days (n=4)
  Arms: Placebo for 1.0 g GLY-200 arm
Drug: Placebo — 4 placebo capsules BID for 14 days (n=4)
  Arms: Placebo for 2.0 GLY-200 arm

SUMMARY:
This study is a Phase 2, randomized, double-blind, placebo-controlled, single-center study in adult patients with type 2 diabetes. It will evaluate the safety and tolerability of oral GLY-200. Subjects will participate in a ≤ 18-day screening period followed by a metformin washout period of approximately 14 days, and an inpatient period of 16 days. Approximately 48 subjects will be randomized to 1 of 3 active treatment groups or 1 of 3 placebo groups. Dosing will occur for 14 days. A follow-up clinic visit will occur on Day 21 [End of Study (EOS)] or Early Termination (ET).

ELIGIBILITY:
Key Inclusion Criteria:

* Patients diagnosed with type 2 diabetes: hemoglobin A1c (HbA1c)) ≥ 6.0 and ≤ 8.5% at screening
* Body mass index (BMI) ≥ 18 and ≤ 40 at screening

Key Exclusion Criteria:

* Treated with any prescription medication for the treatment of type 2 diabetes or weight loss other than metformin in the last 3 months prior to screening
* Use of any drug treatment that affects gastric pH
* Use of any drug treatment that affects gastrointestinal motility
* Fasting blood glucose > 190 mg/dL
* Diagnosis or treatment of any clinically symptomatic biochemical or structural abnormality of the gastrointestinal (GI) tract or active disease within 12 months prior to screening
* History of any previous abdominal or intestinal surgery including endoscopic, open or laparoscopic thoracic or abdominal surgery, surgical resection of the stomach, small or large intestine
* Clinically significant medical condition as judged by the Investigator that could potentially affect study participation and/or personal well-being

Ages: 30 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2022-08-03 (Actual); Primary Completion 2023-03-14 (Actual); Study Completion 2023-03-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Fineman, PhD, Study Chair — Glyscend, Inc.
Locations (1):
- ProSciento, Inc., Chula Vista, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bryant CLN, Colbert K, Hompesch M, Chaves S, Nimgaonkar A, Fineman MS. GLY-200, an oral pharmacologic duodenal exclusion drug, resulted in positive effects on glucose, lipids and bodyweight in patients with type 2 diabetes: Results of a randomized, double-blind placebo-controlled trial. Diabetes Obes Metab. 2025 Oct;27(10):5996-6005. doi: 10.1111/dom.16664. Epub 2025 Aug 6. PMID 40767317

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A metformin washout period was to take place from Day -14 to Day 1 (a total of 14 days).
Groups:
- 0.5 g GLY-200: 0.5 g GLY-200 (1 x 0.5 g capsule) orally twice a day for 14 days
- 1.0 g GLY-200: 1.0 g GLY-200 (2 x 0.5 g capsules) orally twice a day for 14 days
- 2.0 g GLY-200: 2.0 g GLY-200 (4 x 0.5 g capsules) orally twice a day for 14 days
- Pooled Placebo: Subjects who received 1, 2, or 4 capsules of placebo (orally twice a day for 14 days) were pooled together as the placebo treatment group.
Period: Overall Study
Arm/Group | 0.5 g GLY-200 | 1.0 g GLY-200 | 2.0 g GLY-200 | Pooled Placebo
Started | 14 | 12 | 13 | 12
Completed | 12 | 11 | 10 | 11
Not Completed | 2 | 1 | 3 | 1
Not completed — Withdrawal by Subject | 0 | 1 | 2 | 0
Not completed — COVID-19 Infection | 2 | 0 | 1 | 1

BASELINE CHARACTERISTICS:
Population: All randomized participants.
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.5 g GLY-200 | 1.0 g GLY-200 | 2.0 g GLY-200 | Pooled Placebo | Total
Number analyzed (Participants) | 14 | 12 | 13 | 12 | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 56.8 (8.74) | 52.5 (7.29) | 58.1 (7.72) | 57.6 (7.99) | 56.3 (8.04)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 5 | 5 | 3 | 22
  Male | 5 | 7 | 8 | 9 | 29
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10 | 10 | 9 | 9 | 38
  Not Hispanic or Latino | 4 | 2 | 4 | 3 | 13
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 1 | 0 | 0 | 0 | 1
  Black or African American | 1 | 0 | 1 | 2 | 4
  White | 8 | 11 | 12 | 9 | 40
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 0 | 1 | 5
Region of Enrollment [Number; unit: participants]
  United States | 14 | 12 | 13 | 12 | 51
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 29.84 (4.624) | 32.04 (4.849) | 31.82 (4.094) | 31.68 (3.168) | 31.29 (4.219)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events [Safety and Tolerability of GLY-200]
Description: Safety and tolerability will be assessed by incidence of adverse events (AEs). Clinically significant changes from baseline in vital signs, clinical laboratory parameters, and electrocardiograms (ECGs) will be recorded as AEs.
Time Frame: Over the 14-day treatment period
Population: Safety Analysis Set
Measure: Count of Participants; unit: Participants
Arm/Group | 0.5 g GLY-200 | 1.0 g GLY-200 | 2.0 g GLY-200 | Pooled Placebo
Number analyzed (Participants) | 14 | 12 | 13 | 12
Participants | 9 | 8 | 12 | 7

2. Secondary Outcome: Change From Baseline in Fasting Glucose
Description: Evaluate change from baseline (Day 1) in fasting glucose as captured via continuous glucose monitoring (CGM) at Week 1 and Week 2
Time Frame: Day 1, Day 7, and Day 14
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | 0.5 g GLY-200 | 1.0 g GLY-200 | 2.0 g GLY-200 | Pooled Placebo
Number analyzed (Participants) | 14 | 12 | 13 | 12
mg/dL
  Change from Day 1 at Week 1 | -10.04 (27.966) | -5.68 (23.202) | -15.61 (34.160) | 4.86 (22.160)
  Change from Day 1 at Week 2 | -22.56 (30.842) | -13.23 (25.009) | -14.68 (33.097) | 3.48 (29.071)
Statistical Analysis 1: Comparison: 0.5 g GLY-200 vs Pooled Placebo; Analysis at Week 2; Test type: Superiority; p = 0.0007, ANCOVA; Least Squares (LS) Mean Difference = -35.05, 95% CI 2-sided [-54.35 to -15.75]
Statistical Analysis 2: Comparison: 1.0 g GLY-200 vs Pooled Placebo; Analysis at Week 2; Test type: Superiority; p = 0.0193, ANCOVA; LS Mean Difference = -23.14, 95% CI 2-sided [-42.32 to -3.97]
Statistical Analysis 3: Comparison: 2.0 g GLY-200 vs Pooled Placebo; Analysis at Week 2; Test type: Superiority; p = 0.0243, ANCOVA; LS Mean Difference = -21.64, 95% CI 2-sided [-40.33 to -2.96]

3. Secondary Outcome: Change From Baseline in Fasting Plasma Insulin
Description: Evaluate change from baseline in fasting plasma insulin at Day 1, Day 7, and Day 14
Time Frame: Day 1, Day 7, and Day 14
Population: Per Protocol Analysis Set
Measure: Mean (Standard Deviation); unit: mU/L
Arm/Group | 0.5 g GLY-200 | 1.0 g GLY-200 | 2.0 g GLY-200 | Pooled Placebo
Number analyzed (Participants) | 12 | 12 | 10 | 11
mU/L
  Change from Baseline at Day 1 | -0.25 (2.57) | -1.17 (3.15) | 2.03 (3.18) | 1.02 (1.92)
  Change from Baseline at Day 7 | -1.16 (3.36) | -0.76 (3.49) | -1.18 (3.35) | 0.65 (2.84)
  Change from Baseline at Day 14 | -1.11 (3.17) | -0.74 (3.52) | -0.42 (4.49) | 1.19 (2.36)

4. Secondary Outcome: Change From Baseline in 3-hours Postprandial Plasma Glucose Profile
Description: Evaluate change from baseline in Area Under the Curve (AUC) glucose during mixed meal tolerance tests (MMTTs) at Day 1, Day 7, and Day 14. AUC is calculated from -60 to 180 min using the trapezoidal rule.
Time Frame: Day 1, Day 7, and Day 14
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mg/dL*hr
Arm/Group | 0.5 g GLY-200 | 1.0 g GLY-200 | 2.0 g GLY-200 | Pooled Placebo
Number analyzed (Participants) | 14 | 12 | 13 | 12
mg/dL*hr
  Change from baseline absolute AUC at Day 1 | 8.48 (146.856) | -9.30 (91.393) | -17.01 (82.447) | 1.86 (98.33)
  Change from baseline absolute AUC at Day 7 | -79.21 (188.194) | -53.19 (104.891) | -69.05 (126.897) | -2.37 (106.430)
  Change from baseline absolute AUC at Day 14 | -70.47 (280.038) | -66.46 (168.051) | -62.53 (145.027) | 47.16 (124.381)
Statistical Analysis 1: Comparison: 0.5 g GLY-200 vs Pooled Placebo; Analysis at Day 14; Test type: Superiority; p = 0.0298, ANCOVA; LS Mean Difference = -155.68, 95% CI 2-sided [-295.35 to -16.01]
Statistical Analysis 2: Comparison: 1.0 g GLY-200 vs Pooled Placebo; Analysis at Day 14; Test type: Superiority; p = 0.0433, ANCOVA; LS Mean Difference = -143.74, 95% CI 2-sided [-282.92 to -4.55]
Statistical Analysis 3: Comparison: 2.0 g GLY-200 vs Pooled Placebo; Analysis at Day 14; Test type: Superiority; p = 0.0201, ANCOVA; LS Mean Difference = -178.33, 95% CI 2-sided [-327.16 to -29.50]

5. Secondary Outcome: Change From Baseline in 3-hours Postprandial Plasma Insulin Profile
Description: Evaluate change from baseline in Area Under the Curve (AUC) insulin during mixed meal tolerance tests (MMTTs) at Day 1, Day 7, and Day 14. AUC is calculated from -60 to 180 min using the trapezoidal rule.
Time Frame: Day 1, Day 7, and Day 14
Population: Full Analysis Set
Measure: Mean (Standard Deviation); unit: mU/L*hr
Arm/Group | 0.5 g GLY-200 | 1.0 g GLY-200 | 2.0 g GLY-200 | Pooled Placebo
Number analyzed (Participants) | 14 | 12 | 13 | 12
mU/L*hr
  Change from baseline absolute AUC at Day 1 | -19.49 (38.268) | -3.15 (45.187) | -44.18 (77.942) | 6.13 (37.07)
  Change from baseline absolute AUC at Day 7 | -20.75 (50.901) | -20.84 (41.769) | -23.00 (52.366) | 55.72 (198.804)
  Change from baseline absolute AUC at Day 14 | -12.71 (72.558) | -30.11 (54.226) | -10.70 (25.343) | 32.32 (145.992)
Statistical Analysis 1: Comparison: 0.5 g GLY-200 vs Pooled Placebo; Analysis at Day 14; Test type: Superiority; p = 0.1992, ANCOVA; LS Mean Difference = -47.07, 95% CI 2-sided [-119.94 to 25.81]
Statistical Analysis 2: Comparison: 1.0 g GLY-200 vs Pooled Placebo; Analysis at Day 14; Test type: Superiority; p = 0.0617, ANCOVA; LS Mean Difference = -70.32, 95% CI 2-sided [-144.26 to 3.61]
Statistical Analysis 3: Comparison: 2.0 g GLY-200 vs Pooled Placebo; Analysis at Day 14; Test type: Superiority; p = 0.2981, ANCOVA; LS Mean Difference = -39.84, 95% CI 2-sided [-116.22 to 36.53]

ADVERSE EVENTS:
Time Frame: Approximately 2 months
Arm/Group | 0.5 g GLY-200 | 1.0 g GLY-200 | 2.0 g GLY-200 | Pooled Placebo
All-Cause Mortality (participants affected / at risk) | 0/14 | 0/12 | 0/13 | 0/12
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/12 | 0/13 | 0/12
Other Adverse Events (participants affected / at risk) | 9/14 | 8/12 | 12/13 | 7/12
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 0.5 g GLY-200 (N=14) | 1.0 g GLY-200 (N=12) | 2.0 g GLY-200 (N=13) | Pooled Placebo (N=12)
Constipation (Gastrointestinal disorders) | 8 (8) | 2 (2) | 7 (10) | 3 (4)
Diarrhoea (Gastrointestinal disorders) | 1 (1) | 4 (5) | 7 (13) | 2 (2)
Nausea (Gastrointestinal disorders) | 2 (4) | 2 (5) | 9 (69) | 1 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (3) | 5 (11) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 3 (3) | 0 (0)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 0 (0) | 3 (6) | 0 (0)
Coronavirus Infection (Infections and infestations) | 2 (2) | 0 (0) | 1 (1) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 1 (1) | 2 (3) | 0 (0)
Abdominal Discomfort (Gastrointestinal disorders) | 0 (0) | 1 (1) | 3 (3) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 2 (4)
Eructation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (3) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-10-06): https://cdn.clinicaltrials.gov/large-docs/25/NCT05478525/Prot_000.pdf
  • Statistical Analysis Plan (2023-04-12): https://cdn.clinicaltrials.gov/large-docs/25/NCT05478525/SAP_001.pdf